CLINICAL TRIAL: NCT07269223
Title: Effect Of Oral Vitamin D3 Supplementation On Inflammatory Biomarkers In Patients With Ulcerative Colitis
Brief Title: Oral Vitamin D3 Effect on Inflammatory Biomarkers in Ulcerative Colitis Patients
Acronym: OVDIEIBUCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Qaisar Raza, Assistant Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversityUVAS; UVAS (Other: UNIVERSITY OF VETERINARY & ANIMAL SCIENCES, LAHORE)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; Vitamin D; Immune modulation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the treatment group (Vitamin D3 supplementation plus standard care) or the control group (standard care only). Both groups will be followed concurrently for 12 weeks to assess changes in inflammatory biomarkers, disease activity, and vitamin D status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Placebo Comparator): Intervention Type: Drug Intervention Name: Placebo Capsule
  Description:
  "An inactive oral placebo capsule that contains no Vitamin D3. It is matched in appearance and administration schedule to the active supplement and is used to maintain blinding."
  Interventions: Drug: Vitamin D3
- 2 (Experimental): Intervention Type: Drug Intervention Name: Vitamin D3
  Description:
  "This intervention consists of oral Vitamin D3 (cholecalciferol) capsules administered every two weeks to improve vitamin D status. The dose is designed to raise serum 25(OH)D levels. Adherence will be monitored using supplement logs and follow-up visits."
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — This intervention consists of oral Vitamin D3 (cholecalciferol) capsules administered every two weeks for the duration of the study. The dose is designed to raise and maintain adequate serum 25-hydroxyvitamin D levels. Participants will receive the active supplement under supervised distribution, and adherence will be monitored through supplement logs and follow-up visits

SUMMARY:
This randomized controlled trial aims to evaluate the effect of oral vitamin D3 supplementation on inflammatory biomarkers and disease activity in Pakistani patients with moderate ulcerative colitis. Sixty patients will be randomized to receive either standard treatment alone/Placebo or standard treatment plus vitamin D3 (50,000 IU fortnightly) for 12 weeks. Primary outcomes include changes in blood (CRP, ESR, IL-6) and fecal (calprotectin) inflammatory biomarkers, and disease activity assessed by the partial Mayo score. Secondary outcomes include vitamin D status, dietary intake, and quality of life. The study will provide insights into the immune-modulating and anti-inflammatory role of vitamin D3 as an adjunct therapy in ulcerative colitis.

DETAILED DESCRIPTION:
Background: Ulcerative colitis is a subtype of inflammatory bowel disease that affects the colon and is characterized by alternating phases of relapse (active disease) and remission (normal state). It results in bloody diarrhea and frequent bowel movement. An abnormal mucosal immune response arising from intolerance towards luminal antigens is a hallmark of ulcerative colitis. Vitamin D deficiency is highly prevalent in ulcerative colitis patients. Vitamin D3 improves exaggerated immune responses by increasing the number of Treg cells, suppressing the activity of Th1/Th17 cells (modulating pro-inflammatory cytokine). Thus, it reduces inflammation, neutrophils migration towards mucosa and improves intestinal epithelial barrier function. It also enhances the response of medicines. There is a lack of interventional studies evaluating the anti-inflammatory and immune-modulating role of vitamin D3 in severely vitamin D deficient patients with ulcerative colitis. The current study aims to assess the effect of oral vitamin D3 supplementation on serum and fecal inflammatory biomarkers, and disease activity in moderate ulcerative colitis patients from Pakistani population. This study will help to reduce disease symptoms and improve quality of life of ulcerative colitis patients.

Hypothesis: Oral vitamin D3 supplementation is effective to improve blood and fecal inflammatory biomarkers in Pakistani patients with moderate ulcerative colitis Objectives i. To assess the effect of oral vitamin D3 supplementation on blood and fecal inflammatory biomarkers (i.e., ESR, CRP, IL-6, and calprotectin) in Pakistani patients with moderate ulcerative colitis ii. To evaluate the impact of oral vitamin D3 supplementation on disease activity in Pakistani patients with moderate ulcerative colitis using the partial Mayo score iii. To determine the risk of vitamin D deficiency in Pakistani patients with moderate ulcerative colitis using 24-hour dietary recalls Methodology: It will be a randomized controlled trial. The participants meeting study inclusion criteria will be enrolled. Total sixty (n=60) patients with moderately active condition ulcerative colitis (based on standard clinical i.e Truelove and Witts and colonoscopic criteria) will be recruited from the Department Gastroenterology and Hepatology, Sheikh Zayed Hospital, Lahore. The duration of this clinical will be 12 weeks. Both male and female patients will be included and any patient who has taken vitamin D supplements within three months prior to the study will be excluded. Convenient sampling technique will be used to obtain data. All the participants will be divided into 2 groups: Control group and Treatment group. The control group will be asked to take their medicines only as prescribed by physician and will also be given placebo. Meanwhile, patients in the treatment group will be provided with vitamin D3 capsules (50,000 IU) and advised to consume one capsule after every two weeks (fortnightly) in addition to their medicines. The drug type and its dosage will remain same throughout clinical trial in both groups. The baseline data will comprise of demographic profile, disease duration, blood inflammatory biomarker i.e CRP, ESR, and IL-6, fecal biomarker i.e calprotectin, anthropometric measurements (weight, height, BMI), Vitamin D status. Two 24-hour dietary recalls on two non-consecutive days will also be taken before and after the study. Data regarding stool frequency and blood in stool, and physician's assessment to calculate partial Mayo score will also be collected. Patient follow-up will be conducted through phone calls and in-person meetings. After 12 weeks, the same protocol as the baseline visit (excluding the demographic profile) will be followed.

Statistical Analysis Data will be analyzed through SPSS version 25.0. Results will be presented in the form of descriptive and inferential statistics. Quantitative variables like weight, ESR, CRP, IL-6, fecal calprotectin, vitamin D status and BMI will be reported by mean ± standard deviation. In addition, gender and study groups will be assessed by using frequency and percentages. Baseline and post-study results (before and after) of every group will be compared by paired sample t-test. Results of both groups will be compared by independent sample t-test. Results of drugs-based subgroups will be compared by using one-way ANOVA. P-value ≤ 0.05 will be considered significant. Multiple logistic regression analysis will be used to control for confounding variables in the 24-hour dietary recall data.

Expected Outcomes The current study will provide valuable insights regarding the beneficial role of vitamin D3. Oral vitamin D3 may improve inflammatory biomarkers, reduces disease activity, corrects vitamin D deficiency, and enhance drug response in Pakistani patients with moderate ulcerative colitis, supporting its role as a safe and cost-effective adjunct therapy. Thus, it is expected that patient's disease symptoms and quality of life will be improved.

ELIGIBILITY:
Inclusion Criteria:

* • All patients diagnosed previously by standard clinical i.e Truelove and Witts and endoscopic/ colonoscopic criteria

  * Patients with moderate ulcerative colitis will be included
  * Both male and female patients will be included in the study
  * No change in the type and dosage of their medicine over the past month
  * Patient with severe vitamin D deficiency (< 10 ng/mL) after screening
  * Patients who will provide written informed consent
  * Age: 20-40 year

Exclusion Criteria:• Patients using Vitamin D supplement in the 3 months before the study

* Patients suffering from Crohn's disease or any known autoimmune disease
* Patients with mild and severe ulcerative colitis
* Changes in the type and dosage of the drug during the study
* Pregnant and lactating women
* Patients with known kidney disease
* Patients with known liver disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Name: Change in ESR Unit: mm/hr | Baseline and week 12
  Standard Westergren method
Name: Change in CRP Unit: mg/L | Baseline to 12 weeks
  Measured by immunoturbidimetry
Name: Change in serum IL-6 Unit: pg/mL | Baseline to 12 weeks
  Measured using ELISA
Change in fecal calprotectin concentration Unit: µg/g | Baseline and 12 weeks
  Fecal calprotectin measured using quantitative ELISA.

SECONDARY OUTCOMES:
Name: Change in serum 25-hydroxyvitamin D (25-OH Vitamin D) levels Unit: ng/mL | Baseline and 12 weeks
  Serum 25-OH Vitamin D levels will be measured using chemiluminescent immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Qaisar Raza, PhD, Principal Investigator — UNIVERSITY OF VETERINARY & ANIMAL SCIENCES, LAHORE
Locations (1):
- University of Veterinary & Animal Sciences, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No